CLINICAL TRIAL: NCT00234689
Title: Efficacy of Naltrexone Treatment as Augmentation to SSRI in OCD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Joseph Zohar, Chaim Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SHEBA-99-1897-JZ-CTIL
Record Dates: First submitted 2005-10-06; First posted 2005-10-07 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
Assessing the efficacy of Naltrexone as augmentation to SSRI in patients with OCD

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD
* Treatment with SSRI for at least 10 weeks with no response

Exclusion Criteria:

* Suffering from any medical condition
* treatment with opiates
* chronic use of drugs
* Hepatitis or other liver related diseases
* Incapability to sign an informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, MD, Principal Investigator — Tel Aviv University; Revital Amiaz, MD, Study Chair — Tel Aviv University
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel